CLINICAL TRIAL: NCT03802526
Title: Pharmacokinetic Interaction and Safety/Tolerability Between NVP-1805-R1 and NVP-1805-R2 in Healthy Volunteers
Brief Title: Pharmacokinetic Interaction and Safety/Tolerability Between NVP-1805-R1 and NVP-1805-R2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1805_DDI
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NVP-1805-R1 (Experimental): Drug: NVP-1805-R1
  1 tablet, oral dosing
  Interventions: Drug: NVP-1805-R1
- NVP-1805-R2 (Experimental): Drug: NVP-1805-R2
  1 tablet, oral dosing
  Interventions: Drug: NVP-1805-R2
- NVP-1805-R1 and NVP-1805-R2 (Experimental): Drug: NVP-1801-R1 1 tablet and NVP-1801-R2 1 tablet co-administration(oral dosing)
  Interventions: Drug: NVP-1805-R1 and NVP-1805-R2

INTERVENTIONS:
Drug: NVP-1805-R1 — 1 tablet, multiple oral dosing
  Other Names: NVP-1805-R1(M)
  Arms: NVP-1805-R1
Drug: NVP-1805-R2 — 1 tablet, multiple oral dosing
  Other Names: NVP-1805-R2(C)
  Arms: NVP-1805-R2
Drug: NVP-1805-R1 and NVP-1805-R2 — NVP-1805-R1,1 tablet and NVP-1805-R2, 1 tablet, co-administration, multiple oral dosing
  Other Names: NVP-1805-R1(M) and NVP-1805-R2(C)
  Arms: NVP-1805-R1 and NVP-1805-R2

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and safety/tolerability between NVP-1805-R1 and NVP-1805-R2

DETAILED DESCRIPTION:
pharmacokinetics and safety/tolerability between NVP-1805-R1 and NVP-1805-R2

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 19-45 years.
* BMI of >18.5 kg/㎡ and <27.0 kg/㎡ subject, weight more than 50kg.
* Voluntarily provided a witten consent to participate in this clinical study.

Exclusion Criteria:

* Treatment with an investigational product (Phase I study or Biological study) within 3month preceeding the first dose of study medication.
* History of (or presence) study medication absortion, distribution, metabolism(e.g., liver/ductal, kidney, cardio-vascular, endocrine, respiratory, GI, hematology, oncology, CNS, musculo-skeletal) or related past medical/surgery history
* Pregnant or lactating women.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic interaction | 0hours - 48hours
  Area under the curve (AUC)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Sung Shin, M.D., Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim CH, Kang SI, Shin D. Pharmacokinetic Interaction Between Telmisartan and Rosuvastatin/Ezetimibe After Multiple Oral Administration in Healthy Subjects. Adv Ther. 2021 Feb;38(2):1094-1105. doi: 10.1007/s12325-020-01592-8. Epub 2020 Dec 16. PMID 33326064